CLINICAL TRIAL: NCT01619839
Title: A Phase 2, Enriched-Enrollment, Randomized-Withdrawal, Double-Blind, Placebo-Controlled, Multi-Center Study to Assess the Efficacy, Tolerability, and Safety of NKTR-181 in Opioid-Naïve Subjects With Moderate to Severe Chronic Pain Due to Osteoarthritis of the Knee
Brief Title: A Phase 2 Study To Assess The Efficacy, Tolerability, And Safety OF NKTR-181 In Subjects With Chronic OA Knee Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-181-04
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Results first posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Osteoarthritis of the Knee
Keywords: Nektar; NKTR-181
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — NKTR-181

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 100 mg NKTR-181 (Experimental): 100 mg of NKTR-181 in tablet form, BID. Dosing to occur at Titration period up to 30 days and at Randomization period up to 24 days.
  Interventions: Drug: NKTR-181
- 200 mg NKTR-181 (Experimental): 200 mg of NKTR-181 in tablet form, BID. Dosing to occur at Titration period up to 30 days and at Randomization period up to 24 days.
  Interventions: Drug: NKTR-181
- 300 mg NKTR-181 (Experimental): 300 mg of NKTR-181 in tablet form, BID. Dosing to occur at Titration period up to 30 days and at Randomization period up to 24 days
  Interventions: Drug: NKTR-181
- 400 mg NKTR-181 (Experimental): 400 mg of NKTR-181 in tablet form, BID. Dosing to occur at Titration period up to 30 days and at Randomization period up to 24 days
  Interventions: Drug: NKTR-181
- Placebo (Placebo Comparator): Placebo dosing will be only in the double-blind randomization arm and will be identical in form to the Experimental NKTR-181.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NKTR-181
  Arms: 100 mg NKTR-181; 200 mg NKTR-181; 300 mg NKTR-181; 400 mg NKTR-181
Drug: Placebo — Placebo dosing will be only in the double-blind randomization arm and will be identical in form to the Experimental NKTR-181
  Arms: Placebo

SUMMARY:
NKTR-181 is being developed as an analgesic compound for the treatment of moderate to severe chronic pain - active as a mu agonist, but with inherent molecular properties designed to provide a unique clinical profile, including most notably, reduced CNS side effects and an attenuated attractiveness as a target of abuse.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent;
* Willing and able to understand the study procedures, and comply with all study procedures;
* Females or males, age ≥ 18 years old;
* Body mass index 18-39, inclusive;
* In good general health;
* Clinical diagnosis of OA in one or both knees;
* Have been on a stable regimen of pain medication for the management of OA knee pain;
* Not experiencing adequate pain relief with their current dosing regimen;
* Women of childbearing potential (WCBP) must agree to use highly effective methods of birth control. Male subjects must agree to use contraception.

Exclusion Criteria:

* Females who are pregnant or lactating;
* Known history of hypersensitivity, intolerance, or allergy to opioids;
* Diagnosed as having any chronic pain symptom that in the Investigator's opinion would interfere with the assessment of pain and other symptoms of OA;
* Presence of any medical condition that would preclude study participation in the opinion of the investigator;
* Clinically significant abnormalities of vital signs or clinical laboratory results;
* Clinically significant electrocardiographic abnormalities;
* Received systemic corticosteroids within 30 days prior to signing the consent form;
* Subjects who are known or suspected to be currently abusing alcohol or drugs;
* Positive urine drug screen, or alcohol breath test during Screening Period testing;
* Positive serology for the surface antigen of Hepatitis B (HBsAg) or Hepatitis C (anti-HCV) during Screening Period testing;
* Known to be human immunodeficiency virus (HIV) positive;
* Donation of blood or plasma within 30 days prior to signing the consent form;
* Participation in another drug or biologic study within 30 days prior to signing the consent form;
* Any other reason that, in the opinion of the Investigator or Medical Monitor, would render the subject unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2012-06; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Nektar Therapeutics
Locations (32):
- United States (32):
  - Investigator Site - Mobile, Mobile, Alabama
  - Investigator Site - Tuscon, Tucson, Arizona
  - Investigator Site - Garden Grove, Garden Grove, California
  - Investigator Site - San Diego, San Diego, California
  - Investigator Site - Walnut Creek, Walnut Creek, California
  - Investigator Site - Westlake Village, Westlake Village, California
  - Investigator Site - Coral Gables, Coral Gables, Florida
  - Investigator Site - Fort Meyers, Fort Myers, Florida
  - Investigator Site - Pembroke Pines, Pembroke Pines, Florida
  - Investigator Site - West Palm Beach, West Palm Beach, Florida
  - Investigator Site - Weston, Weston, Florida
  - Investigator Site - Evansville, Evansville, Indiana
  - Investigator Site - Wichita, Wichita, Kansas
  - Investigator Site - Louisville, Louisville, Kentucky
  - Investigator Site - Brockton, Brockton, Massachusetts
  - Investigator Site - Worcester, Worcester, Massachusetts
  - Investigator Site - Kansas City, Kansas City, Missouri
  - Investigator Site - Omaha, Omaha, Nebraska
  - Investigator Site - Las Vegas, Las Vegas, Nevada
  - Investigator Site - Berlin, Berlin, New Jersey
  - Investigator Site - Englewood, Englewood, New Jersey
  - Investigator Site - Greensboro, Greensboro, North Carolina
  - Investigator Site - Cincinnati, Cincinnati, Ohio
  - Investigator Site - Oklahoma City, Oklahoma City, Oklahoma
  - Investigator Site - Duncansville, Duncansville, Pennsylvania
  - Investigator Site - Philadelphia, Philadelphia, Pennsylvania
  - Investigator Site - Charleston, Charleston, South Carolina
  - Investigator Site - Austin, Austin, Texas
  - Investigator Site - Dallas, Dallas, Texas
  - Investigator Site - San Antonio, San Antonio, Texas
  - Investigator Site - Salt Lake City, Salt Lake City, Utah
  - Investigator Site - Kenosha, Kenosha, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 296 subjects were enrolled in this study. Of these, one subject did not receive study drug in the open-label Titration Period because she had a history of drug abuse and thus did not meet entry criteria. Of the 295 subjects dosed during the open-label Titration Period, 213 subjects were randomized to treatment. All 295 subjects who received study drug were included in the safety analysis population.
Groups:
- 100 mg NKTR-181: 100 mg of NKTR-181 in tablet form, BID. Dosing to occur at Titration period up to 30 days and at Randomization period up to 24 days.
  NKTR-181
- 200 mg NKTR-181: 200 mg of NKTR-181 in tablet form, BID. Dosing to occur at Titration period up to 30 days and at Randomization period up to 24 days.
  NKTR-181
- 300 mg NKTR-181: 300 mg of NKTR-181 in tablet form, BID. Dosing to occur at Titration period up to 30 days and at Randomization period up to 24 days
  NKTR-181
- 400 mg NKTR-181: 400 mg of NKTR-181 in tablet form, BID. Dosing to occur at Titration period up to 30 days and at Randomization period up to 24 days
  NKTR-181
Period: Overall Study
Arm/Group | 100 mg NKTR-181 | 200 mg NKTR-181 | 300 mg NKTR-181 | 400 mg NKTR-181 | Placebo
Started | 48 | 31 | 18 | 10 | 106
Completed | 43 | 27 | 17 | 9 | 97
Not Completed | 5 | 4 | 1 | 1 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 100 mg NKTR-181 | 200 mg NKTR-181 | 300 mg NKTR-181 | 400 mg NKTR-181 | Placebo | Total
Number analyzed (Participants) | 48 | 31 | 18 | 10 | 106 | 213
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (9.77) | 57.6 (11.43) | 60.6 (9.57) | 59.8 (9.51) | 60.1 (9.55) | 60.1 (9.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 18 | 9 | 7 | 66 | 127
  Male | 21 | 13 | 9 | 3 | 40 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 4 | 3 | 21 | 41
  Not Hispanic or Latino | 40 | 25 | 14 | 7 | 83 | 169
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 0 | 1 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 10 | 2 | 1 | 20 | 40
  White | 39 | 19 | 16 | 8 | 82 | 164
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: centimeters] | 170.1 (10.84) | 169.5 (11.55) | 169.7 (9.41) | 168.0 (11.37) | 167.2 (10.40) | 168.4 (10.62)
Weight [Mean (Standard Deviation); unit: kilograms] | 89.27 (17.496) | 90.75 (22.355) | 85.85 (16.739) | 84.27 (18.918) | 89.57 (19.116) | 89.11 (18.967)

OUTCOME MEASURES:

1. Primary Outcome: The Mean Change From Baseline Pain Score to Pain Score at the End of the Double-blind Randomized Treatment Period.
Description: The first phase of this trial involved an open-label titration period where patients were given NKTR-181 at increasing doses up to a maximum of 400 mg twice daily until adequate pain control was achieved. Patients achieving adequate pain control were then progressed to the second phase of the trial where patients were randomized in a 1:1 ratio to receive either placebo or their tolerable dose level of NKTR-181.
  All efficacy data for NKTR-181 patients was combined into one group regardless of tolerable dose level. For this outcome, the subjects had to rate their worst pain intensity during the past 4 hours from 0 to 10 on an 11-point scale, where 0 represented one end of the continuum (i.e., no pain) and 10 represented the other extreme of pain intensity (i.e., worst pain imaginable).
Time Frame: Baseline and Visit 10 (day 69)
Measure: Mean (Standard Error); unit: Change in Pain Score
Groups:
- NKTR-181: Patients who received at least one dose of NKTR-181
- Placebo: Patients given placebo
Arm/Group | NKTR-181 | Placebo
Number analyzed (Participants) | 106 | 106
Change in Pain Score | -0.06 (0.162) | -0.01 (0.168)

2. Secondary Outcome: Time to Discontinuation During the Double-blind Randomized Treatment Period for Any Reason
Description: The first phase of this trial involved an open-label titration period where patients were given NKTR-181 at increasing doses up to a maximum of 400 mg twice daily until adequate pain control was achieved. Patients achieving adequate pain control were then progressed to the second phase of the trial where patients were randomized in a 1:1 ratio to receive either placebo or their tolerable dose level of NKTR-181.
  All efficacy data for NKTR-181 patients was combined into one group regardless of tolerable dose level.
Time Frame: Randomization Treatment period is 24 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | NKTR-181 | Placebo
Number analyzed (Participants) | 106 | 106
days | 20.2 (4.21) | 20.2 (3.86)

ADVERSE EVENTS:
Description: Please note that the number of participants at risk analyzed for Serious Adverse Events includes all patients that were enrolled in the study not just the ones that were randomized to treatment.
Arm/Group | 100 mg NKTR-181 | 200 mg NKTR-181 | 300 mg NKTR-181 | 400 mg NKTR-181 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/31 | 0/18 | 0/10 | 0/106
Serious Adverse Events (participants affected / at risk) | 0/133 | 1/84 | 0/46 | 1/32 | 0/0
Other Adverse Events (participants affected / at risk) | 27/48 | 19/31 | 11/18 | 5/10 | 54/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 100 mg NKTR-181 (N=133) | 200 mg NKTR-181 (N=84) | 300 mg NKTR-181 (N=46) | 400 mg NKTR-181 (N=32) | Placebo (N=0)
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Coronary Artery Stenosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 100 mg NKTR-181 (N=48) | 200 mg NKTR-181 (N=31) | 300 mg NKTR-181 (N=18) | 400 mg NKTR-181 (N=10) | Placebo (N=106)
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1
Lacrimation Increased (Eye disorders) | 0 | 0 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 9 | 8 | 5 | 2 | 15
Nausea (Gastrointestinal disorders) | 4 | 4 | 3 | 0 | 7
Dry Mouth (Gastrointestinal disorders) | 2 | 2 | 1 | 0 | 3
Vomiting (Gastrointestinal disorders) | 1 | 4 | 0 | 0 | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 5
Fatigue (General disorders) | 1 | 0 | 1 | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 1 | 0 | 4
Gingival Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 2
Somnolence (Nervous system disorders) | 2 | 4 | 0 | 1 | 5
Dizziness (Nervous system disorders) | 2 | 2 | 2 | 0 | 2
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 3 | 0 | 0 | 4
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Heat Exhaustion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There are restrictions to the PI's rights to discuss or publish trial results.